CLINICAL TRIAL: NCT02998372
Title: Computational Simulation of Dynamic Motion for Knees With Patellar Instability to Compare MPFL Reconstruction to Tibial Tuberosity Medialization as a Function of Knee Anatomy
Brief Title: Computational Simulation of Patellar Instability
Status: Terminated | Type: Observational
Why Stopped: Not reaching targeted enrollment
Sponsor: Cleveland Clinic Akron General (Other)
Collaborators: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, John Elias, PhD, Senior Research Scientist, Cleveland Clinic Akron General
Other Study IDs: 110908
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Patellar Instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: patellar stabilization — surgery to either alter soft tissues around the patella or reorient the patellar tendon to restore patellar stability

SUMMARY:
Computational simulation will be performed to represent motion of knees with a dislocating kneecap. Common surgical treatment methods will be simulated and anatomical parameters commonly associated with the dislocation will be varied in order to characterize the most appropriate surgical approach as a function of knee anatomy.

DETAILED DESCRIPTION:
The two most common stabilization procedures for patients with recurrent patellar instability are reconstruction of the medial patellofemoral ligament (MPFL) and medialization of the tibial tuberosity. MPFL reconstruction has been growing in popularity, due in large part to the technical demands of tibial tuberosity realignment and concerns related to bone healing across the osteotomy. In cases of severe trochlear dysplasia and/or a dramatically lateralized tibial tuberosity, an MPFL graft tensioned according to current standards may not provide sufficient resistance to limit lateral patellar tracking that causes continued instability. Increasing graft tension could overload medial patellofemoral cartilage. The proposed study is based on the hypothesis that the ability of MPFL reconstruction to effectively limit lateral patellar maltracking decreases as trochlear dysplasia and the lateral position of the tibial tuberosity increase. Computational dynamic simulation of knee function will be performed to establish anatomical standards for which tibial tuberosity medicalization is more likely than MPFL reconstruction to limit patellar maltracking without overloading patellofemoral cartilage. The first specific aim is to computationally replicate lateral patellar maltracking and pressure applied to cartilage during function for patients being treated for patellar instability. Multibody dynamics knee models representing patients being treated for recurrent patellar instability will be based on 3D reconstructions from MRI scans. The modeling technique treats the bones and cartilage surfaces as rigid bodies with Hertzian contact determining contact forces and guiding joint motion. Discrete element analysis techniques will be used to characterize contact pressure patterns based on overlap of cartilage surfaces. Models will be individually validated by comparing output to in vivo data. The source of the in vivo data will be computational reconstruction of in vivo function based on motions performed by the patients who provide the imaging data for model development. The second specific aim will be to computationally characterize the influence of surgical stabilization on knee function for individual patients. MPFL reconstruction and tibial tuberosity medialization, each with variations in surgical parameters, will be simulated. The actual surgical procedures performed on the patients will be simulated, with the influence on lateral tracking compared to in vivo results to validate the representation of the surgical procedures. The third specific aim will be to compare surgical options as a function of patellofemoral anatomy. Variations in patellar tracking and pressure applied to cartilage will be compared between MPFL reconstruction and tuberosity medialization. In addition, techniques to parametrically alter trochlear dysplasia and tuberosity lateralization within the models will be developed. Simulations will be performed while varying anatomy to set ranges over which each surgical option can limit patellar maltracking without elevating contact pressures. The modeling system will be available for future studies addressing additional surgical options and anatomical parameters related to patellar instability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent patellar dislocation
* Plan to be surgically treated at Akron Children's Hospital

Exclusion Criteria:

* Additional Injuries unrelated to patellar instability for the knee of interest
* Implantation of metallic hardware that could cause artifacts within MRI scans
* Inability to remain still during MRI scans

Max Age: 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anyone with a diagnosis of recurrent patellar dislocation to be surgically treated at Akron Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Graphical representation of changes in knee motion due to surgery | 16 months
  Computational models will be developed from MRI scans to show pre-operative and post-operative motion patterns for knees with instability
Computational simulation of changes in knee motion due to surgery | 24 months
  The models used to display motion will be converted to dynamic simulation models to predict the influence of multiple surgical approaches on knee motion

SECONDARY OUTCOMES:
Influence of anatomy on surgical effectiveness | 24 months
  The simulation models will be used to relate the effectiveness of each procedure to the anatomy of the knees

CONTACTS AND LOCATIONS:
Overall Officials: John Elias, PhD, Principal Investigator — Cleveland Clinic Akron General
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elias JJ, Cosgarea AJ. Technical errors during medial patellofemoral ligament reconstruction could overload medial patellofemoral cartilage: a computational analysis. Am J Sports Med. 2006 Sep;34(9):1478-85. doi: 10.1177/0363546506287486. Epub 2006 May 9. PMID 16685097
- [Background] Biyani R, Elias JJ, Saranathan A, Feng H, Guseila LM, Morscher MA, Jones KC. Anatomical factors influencing patellar tracking in the unstable patellofemoral joint. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2334-41. doi: 10.1007/s00167-014-3195-y. Epub 2014 Jul 26. PMID 25063490
- [Background] Elias JJ, Carrino JA, Saranathan A, Guseila LM, Tanaka MJ, Cosgarea AJ. Variations in kinematics and function following patellar stabilization including tibial tuberosity realignment. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2350-6. doi: 10.1007/s00167-014-2905-9. Epub 2014 Feb 15. PMID 24531362
- [Background] Purevsuren T, Elias JJ, Kim K, Kim YH. Dynamic simulation of tibial tuberosity realignment: model evaluation. Comput Methods Biomech Biomed Engin. 2015;18(14):1606-10. doi: 10.1080/10255842.2014.936857. Epub 2014 Jul 15. PMID 25025488
- [Background] Fitzpatrick CK, Steensen RN, Tumuluri A, Trinh T, Bentley J, Rullkoetter PJ. Computational analysis of factors contributing to patellar dislocation. J Orthop Res. 2016 Mar;34(3):444-53. doi: 10.1002/jor.23041. Epub 2015 Sep 15. PMID 26331373
- [Background] Elias JJ, Saranathan A. Discrete element analysis for characterizing the patellofemoral pressure distribution: model evaluation. J Biomech Eng. 2013 Aug;135(8):81011. doi: 10.1115/1.4024287. PMID 23719962
- [Background] Guess TM, Liu H, Bhashyam S, Thiagarajan G. A multibody knee model with discrete cartilage prediction of tibio-femoral contact mechanics. Comput Methods Biomech Biomed Engin. 2013;16(3):256-70. doi: 10.1080/10255842.2011.617004. Epub 2011 Oct 4. PMID 21970765
- [Background] Guess TM, Thiagarajan G, Kia M, Mishra M. A subject specific multibody model of the knee with menisci. Med Eng Phys. 2010 Jun;32(5):505-15. doi: 10.1016/j.medengphy.2010.02.020. Epub 2010 Mar 31. PMID 20359933
- [Background] Elias JJ, Kelly MJ, Smith KE, Gall KA, Farr J. Dynamic Simulation of the Effects of Graft Fixation Errors During Medial Patellofemoral Ligament Reconstruction. Orthop J Sports Med. 2016 Sep 20;4(9):2325967116665080. doi: 10.1177/2325967116665080. eCollection 2016 Sep. PMID 27709116
- [Background] Elias JJ, Soehnlen NT, Guseila LM, Cosgarea AJ. Dynamic tracking influenced by anatomy in patellar instability. Knee. 2016 Jun;23(3):450-5. doi: 10.1016/j.knee.2016.01.021. Epub 2016 Feb 26. PMID 26922799

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02998372/Prot_SAP_000.pdf